CLINICAL TRIAL: NCT04355000
Title: Comparative Evaluation of Effectiveness of Hall Technique and Resin Modified Glass Ionomer Cement in Controlling Occlusoproximal Caries in Dentin of Primary Molars in Children : A Randomized Clinical Study
Brief Title: Comparative Evaluation of Effectiveness of Hall Technique and Resin Modified Glass Ionomer Cement in Controlling Occlusoproximal Caries in Primary Molars in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Saurabh@Pedo#PGIDS
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: Dental Caries
Keywords: RMGIC, Hall Technique, Dental caries in primary molars.
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hall Technique (Active Comparator): In Hall Technique, SS Crown will be cemented on primary carious molar which satisfy the inclusion criterion without any carious removal, without any tooth preperation, without any local anaesthesia.
  Interventions: Procedure: Hall technique
- RMGIC restoration (Active Comparator): In RMGIC(Vitremer) filling, carious lesion will be completely removed from primary molars using air rotor and local anaesthesia according to need and filled with vitremer rmgic material.
  Interventions: Procedure: RMGIC restoration

INTERVENTIONS:
Procedure: Hall technique — SS Crown will be cemented on primary carious molar which satisfy the inclusion criterion without any carious removal, without any tooth preperation, without any local anaesthesia.
  Arms: Hall Technique
Procedure: RMGIC restoration — Complete removal of caries and filling will be done with RMGIC material
  Arms: RMGIC restoration

SUMMARY:
•To investigate clinical and radiographic outcomes of Hall Technique and conventional restorative care using RMGIC in occulusoproximal carious lesions of primary molars in children.

DETAILED DESCRIPTION:
Dental caries is one of the most common preventable diseases which is recognized as the primary cause of oral pain and tooth loss. WHO claimed that poor oral health may have a profound effect on general health as well as quality of life. Dental caries is not an infectious disease that needs to be "cured" by removing bacteria or, even less so, a particular bacterial species. Instead, dental caries can be managed behaviorally by controlling its causative factors-namely, the supply of fermentable carbohydrates and the presence and maturation of bacterial dental biofilms.

Resin modified Glass ionomer cement (RMGIC) has been used as a material for placement of dental restorations and is known to release fluoride which can help to remineralize carious lesion. RMGIC has excellent compressive and tensile strength compared to water based material, very less sensitive to moisture during initial setting time, excellent bonding with tooth, long working time with rapid set and early strength, have lower modulus of elasticity, twice flexible compared to water based glass ionomers. Chisini et al conducted a systematic review and showed 93.6% success rate of RMGIC, 91.2% for compomer, 79.3% for composite resin in primary teeth restoration.

The Hall Technique (HT) is a method for restoring children's carious primary molars uses a preformed stainless steel crown (SSC) cemented with no caries removal, tooth preparation, or local anaesthesia. Schwendicke F reported that HT showed high cost-effectiveness, dominating conventional restoration mainly because HT is clinically more successful and result in significantly fewer retreatments. The Hall Technique has been shown to be a durable (being likely to last the lifespan of the primary molar) and economical management option for primary molars with carious lesions, which in addition offers the benefit of full coronal coverage, reducing the risk of future carious lesion development.

The patients will be randomly allocated into two groups:

Group 1 - 45 Teeth will be treated using Hall Technique. Group 2 - 45 Teeth will be treated using resin modified glass ionomer cement(Vitremer).

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 to 8 years.
* Occlusoproximal caries into dentin affecting one or more than one surface,
* Crown is restorable.
* Absence of clinical signs and symptoms
* More than half root remaining.
* No complicating medical history
* Child able to co-operate.
* Parent and child have consented.
* Patient ready for radiographs.

Exclusion Criteria:

* Signs or symptoms of irreversible pulpitis, or dental abscess/fistula.
* Radiographic signs of pulpal involvement, or periradicular pathology.
* Where there is no cooperation as there is a risk of crown aspiration or swallowing.
* Patients at risk of infective endocarditis; immunocompromised children.
* Parents/carers do not give written consent for treatment.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Clinical success | Baseline to 12 months
  Clinical success will be assessed by absence of clinical signs and symptoms

SECONDARY OUTCOMES:
Radiographic success | Baseline to 12 months
  Absence of periapical alterations (radiolucency at furcal or periapical region).

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India